CLINICAL TRIAL: NCT03859752
Title: A Phase 1, Open Label, First-in-human Study of TR1801-ADC, an Antibody Drug Conjugate (ADC), in Patients With Select Solid Tumors Expressing c-Met
Brief Title: TR1801-ADC in Patients With Tumors That Express c-Met
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Financial funds were withdrawn by investors and study was stopped
Sponsor: Open Innovation Partners, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR1801-CL-01
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: antibody-drug conjugate; c-Met; solid tumors; Phase 1

STUDY DESIGN:
Intervention Model Description: Open label, multiple dose, dose-escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TR1801-ADC (Experimental): Humanized anti-c-Met monoclonal antibody conjugated to a cleavable pyrrolobenzodiazepine toxin
  Interventions: Biological: TR1801-ADC

INTERVENTIONS:
Biological: TR1801-ADC — Humanized anti-c-Met monoclonal antibody conjugated to a cleavable pyrrolobenzodiazepine toxin

SUMMARY:
First-in-human, Phase 1 study to assess safety, tolerability, and pharmacokinetics of TR1801-ADC in patients with select solid tumors that express c-Met.

DETAILED DESCRIPTION:
First-in-human, Phase 1, multiple dose-dose escalation study designed to determine safety, tolerability, maximum tolerated dose, and recommended phase 2 dose of TR1801-ADC in patients with select solid tumors that express c-Met. This study will also assess pharmacokinetics (PK), anti-tumor activity, and correlation between clinical outcomes (safety, anti-tumor activity, and PK) and c-Met expression.

ELIGIBILITY:
Inclusion Criteria:

* Compliance with all study procedures and visits to the clinical research site
* Locally advanced or metastatic disease that is not amenable to definitive therapy
* Histologically confirmed diagnosis of a solid tumor which expresses c-Met
* Must have progressed or have been intolerant to all available therapies known to confer clinical benefit appropriate for the patient's tumor type
* Measurable baseline disease as defined by RECIST Version 1.1
* ECOG Performance Status 0-1
* Body weight within 40 and 150 kg
* Clinical laboratory values with the limits as defined by the protocol
* Not pregnant or breast feeding
* Males and women of child-bearing potential must agree to use an effective method of contraception

Exclusion Criteria:

* Any disease or condition that may be considered to pose an increased risk from study treatment or the ability of the patient to participate and comply with study procedures
* Treatment with anti-cancer therapy (including cytotoxic chemotherapy, major surgery, radiation, biologic and investigational agents) within 21 days before first dose of study treatment
* Brain metastases that has not stabilized for at least 28 days after therapy and who have discontinued steroids for <2 weeks
* Unresolved adverse events >= Grade 2 from prior anticancer therapies
* Acute myocardial infarction, cerebral ischemic infarct, or other arterial thrombosis within 6 months of screening for this study.
* Uncontrolled hypertension, unstable angina, or NYHA Class III/IV heart failure
* History of capillary leak syndrome
* Corticosteroid intolerance
* History of anasarca
* Untreated or uncontrolled bacterial, viral or fungal infection
* HIV infection or active infection with hepatitis B or C
* Significant liver disease
* History of alcoholism or current alcoholism
* Signs of significant portal hypertension
* Significant kidney disease within 2 years
* Active or unstable gallstone disease
* Prior treatment with a c-Met targeted agent
* Prior hypersensitivity reaction to treatment with another monoclonal antibody
* QTcF >=470 ms
* Patients may not start any new herbal or dietary supplement within 4 weeks before initiation of study treatment nor while receiving study treatment
* Administration of a live, attenuated vaccine within 28 days before the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize safety of TR1801-ADC in patients with advanced solid tumor malignancies which express c-Met | 4 years
  Number of participants with treatment-related adverse events
Establish maximum tolerated dose | 3.5 years
  Number of participants with protocol-defined dose-limiting toxicity

SECONDARY OUTCOMES:
Evaluate pharmacokinetics of TR1801-ADC | 4 years
  Analyze blood plasma concentrations
Immunogenicity | 4 years
  Assess anti-drug antibodies of TR1801-ADC
Evaluate clinical activity of TR1801-ADC | 5 years
  Assess objective response rate in accordance with Response Evaluation Criteria in Solid Tumors (RECIST V1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Gordon, MD, Study Director — Open Innovation Partners
Locations (4):
- United States (4):
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - John Hopkins - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - University of Washington / Seattle Cancer Care, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No